CLINICAL TRIAL: NCT01489904
Title: Phase 2/3 Application of Botulinum Neurotoxin Type A in Salivary Glands as a Treatment of Chronic Drooling in Patients With Cerebral Palsy: A Controlled Clinical Trial.
Brief Title: Application of Botulinum Toxin Type A in Salivary Glands in the Treatment of Drooling in Patients With Cerebral Palsy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Vall d'Hebron (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Inma Bori i Fortuny, MD, Neurology- Rehabilitation, Hospital Vall d'Hebron
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-021691-28
Record Dates: First submitted 2011-11-29; First posted 2011-12-12 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Sialorrhea; Cerebral Palsy
Keywords: drooling; cerebral palsy
MeSH Terms: conditions — Sialorrhea; Cerebral Palsy | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botulinum Toxin (Experimental): Botulinum Toxin type-A
  Interventions: Biological: BOTULINUM NEUROTOXIN TYPE-A
- Control Treatment (No Intervention): No intervention

INTERVENTIONS:
Biological: BOTULINUM NEUROTOXIN TYPE-A — Botulinum toxin type A / First infiltration: 25U in each salivary gland=100 U in Parotid and submandibular glands. 24 weeks after first infiltration is a Second infiltration with 50U Botulinum toxin type -A 25 U in each salivary gland only in parotid glands.
  Other Names: Botulinum Neurotoxin type -A; BOTOX
  Arms: Botulinum Toxin

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of botulinum toxin-A in salivary glands as a treatment for decrease drooling in patients with cerebral palsy and evaluate the long-term effects and tolerance . To assess whether patients with cerebral palsy have hypersalivation comparing with patients without treatment and healthy volunteers and if botulinum toxin may reduce the volume of drooling without altering the swallowing function.

DETAILED DESCRIPTION:
Patients with cerebral palsy (CP) and other neurological diseases ( Parkinson´s disease (PD), bulbar amyotrophic lateral sclerosis, neurodegenerative diseases, idiopathic hypersalivation, head and neck carcinomas, etc) frequently have lifelong issues with oral motor control that may present as eating, drinking difficulties, drooling and/or speech problems.

Inadequate saliva control occurs in approximately 30% of patients with CP. Drooling usually caused by swallowing dysfunction and can lead to choking, salivary aspiration, pneumonia, chest infections,chronic irritation of the facial skin, and /or dehydration, in some cases the person loss of self esteem and impede community inclusion.

Numerous therapies, anticholinergic medication, surgery, etc, have all been used to reduce drooling with varying side effects and degrees of success, but none with optimal results.

Systemic anticholinergics may reduce salivary secretion but are frequently not tolerated by the patients because they have multiple side effects. Recently Botulinum toxin type A has been used in the treatment of sialorrhea, in clinical studies have found that botulinum toxin type-A may have a good response with fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cerebral palsy ( medical history, neurological examination,magnetic resonance
* Patients with disorders for eating, drinking, pneumonia, irritation of the skin face, social exclusion
* Score of >3 on drooling severity and frequency scale

Exclusion Criteria:

* Patients under 18 years
* Swallowing disorders
* Diagnosis of Myasthenia, Eaton Lambert Syndrome, Amyotrophic lateral Sclerosis or diseases that interfere with the function neuroglandular
* Pregnant or lactating period
* Patients without informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-11; Primary Completion 2011-11 (Actual); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Asses drool quantification pre and post-infiltration in submandibular and parotid glands with BoNT-A | Change from baseline in drooling0,4,8,12,16,20,24 weeks post infiltration/baseline, and again second infiltration only in parotid glands
  Drool quantification using a pre-and post injection "drool rating scale" dental roll weights, drool quotient.
  Safety evaluate. The proportion of patients with a good response according to the criteria, defined response during treatment or follow-up.

SECONDARY OUTCOMES:
Asses at what period of time after infiltration occurs the maximum response in decreased drooling, and whether Botulinum toxin-A reduce the volume of drooling without altering the swallowing function. | every 4 weeks ( after each infiltration)
  Salivary flow expressed in ml/ min evaluated in diferent subtypes of cerebral palsy compared before and after infiltration and compared with control group without infiltration and control group of healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Maria D González Luis/ Inma Bori, MS/MD, Principal Investigator — Hospital Vall d Hebron. Barcelona Spain
Locations (1):
- CEIC Hospital Vall d Hebron, Barcelona, Barcelona, Spain